CLINICAL TRIAL: NCT00779025
Title: A Safety Evaluation of Personal Lubricant Product When Used by Couples in Home-use Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CA-P-6020-1
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2011-05-05 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Coitus
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MINE Alone (Active Comparator): Female Personal Lubricant (PD-F-5254)
  Interventions: Device: PD-F-5254
- YOURS and MINE (Experimental): Male Personal Lubricant (10855-096) used in conjunction with Female Personal Lubricant (PD-F-5254)
  Interventions: Device: PD-F-5254; Device: 10855-096

INTERVENTIONS:
Device: PD-F-5254 — Female Personal Lubricant (MINE)
  Other Names: K-Y
Device: 10855-096 — Male Personal Lubricant (YOURS)
  Other Names: K-Y
  Arms: YOURS and MINE

SUMMARY:
The purpose of this study is to study in couples and to evaluate the safety of personal lubricant products.

DETAILED DESCRIPTION:
Study to evaluate the safety of Class II personal lubricant devices.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy males and females >18 years of age
* In committed heterosexual relationship for >6months
* On acceptable method of birth control

Exclusion Criteria:

* Pregnant or breastfeeding
* Allergy to product ingredients
* Irritation or infection in genital area
* Unstable or uncontrolled medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wanser, Study Director — J&J CPPW
Locations (1):
- Concentrics Center for Research, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study (ITT): The group evaluated was based on intention to treat (ITT).
Period: Overall Study
Arm/Group | Overall Study (ITT)
Started | 82
Completed | 81
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study (ITT)
Number analyzed (Participants) | 82
Age, Customized [Mean (Standard Deviation); unit: Years]
  Male | 42.3 (14.5)
  Female | 40.0 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Showing Change From Baseline in Irritation Scores
Description: Number of participants showing change in irritation scores based on physical examinations of both male and female subjects according to a 6-point scale, ranging from 0=Normal appearance, no irritation to 6 = Presence of Lesions
Time Frame: 1 week
Population: Analysis was per Intention to Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | MINE Alone | YOURS and MINE
Number analyzed (Participants) | 42 | 40
Participants | 0 (0) | 0 (0)

2. Secondary Outcome: Number of Sensations Experienced by Male Subjects - Overall
Description: Number of sensations experienced by male subjects, based on two applications of the investigational product.
Time Frame: 1 Week
Measure: Number; unit: Sensations
Units Other Than Participants: Applications
Arm/Group | MINE Alone | YOURS and MINE
Number analyzed (Participants) | 21 | 20
Number analyzed (Applications) | 42 | 40
Sensations
  Itching | 0 | 0
  Burning | 2 | 0
  Stinging | 2 | 3
  Tingling | 16 | 15
  Warming | 22 | 24

3. Secondary Outcome: Number of Sensations Experienced by Female Subjects - Overall
Description: Number of sensations experienced by female subjects, based on two applications of the product for each subject.
Time Frame: 1 Week
Population: Intention to Treat
Measure: Number; unit: Sensations
Units Other Than Participants: Applications
Arm/Group | MINE Alone | YOURS and MINE
Number analyzed (Participants) | 21 | 20
Number analyzed (Applications) | 42 | 40
Sensations
  Itching | 1 | 0
  Burning | 4 | 6
  Stinging | 4 | 0
  Tingling | 25 | 22
  Warming | 31 | 22

ADVERSE EVENTS:
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No